CLINICAL TRIAL: NCT06185608
Title: The Effects of Various Concentrations of Ropivacaine on the Onset and Duration of Ultrasound-guided Ankle Blocks in Patients Undergoing Hallux Valgus Repair Surgery - a Randomized, Double-blinded, Parallel-group Interventional Study
Brief Title: The Effects of Various Concentrations of Ropivacaine on the Onset and Duration of Ankle Blocks
Acronym: ROADS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Imré Van Herreweghe, Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROADS
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hallux Valgus; Anesthesia
Keywords: Ropivacaine; Peripheral Nerve Block; Locoregional anesthesia; Onset; Duration; Sensory block
MeSH Terms: conditions — Hallux Valgus | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Staff performing perineural blocks will not be blinded to the concentration of ropivacaine that will be administered. However, patients, and research personnel collecting postoperative data will be blinded to group allocation. The clinical anesthesiologist in the operating theatre is blinded to the concentration of ropivacaine administered as this is not the same practitioner as the one performing the ankle block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0.25% ropivacaine group (Active Comparator): This group will receive a total of 15 mL of 0.25% ropivacaine.
  Interventions: Drug: 0.25% ropivacaine
- 0.5% ropivacaine group (Active Comparator): This group will receive a total of 15 mL of 0.5% ropivacaine.
  Interventions: Drug: 0.5% ropivacaine
- 1% ropivacaine group (Active Comparator): This group will receive a total of 15 mL of 1% ropivacaine.
  Interventions: Drug: 1% ropivacaine

INTERVENTIONS:
Drug: 0.25% ropivacaine — A total of 15 ml of 0.25% ropivacaine will be administered and distributed strategically among the specific nerves: 6 ml for the tibial nerve, 3 ml for the deep peroneal nerve, and 2 ml each for the superficial peroneal nerve, saphenous nerve, and sural nerve.
  Other Names: Group 1
  Arms: 0.25% ropivacaine group
Drug: 0.5% ropivacaine — A total of 15 ml of 0.5% ropivacaine will be administered and distributed strategically among the specific nerves: 6 ml for the tibial nerve, 3 ml for the deep peroneal nerve, and 2 ml each for the superficial peroneal nerve, saphenous nerve, and sural nerve.
  Other Names: Group 2
  Arms: 0.5% ropivacaine group
Drug: 1% ropivacaine — A total of 15 ml of 1% ropivacaine will be administered and distributed strategically among the specific nerves: 6 ml for the tibial nerve, 3 ml for the deep peroneal nerve, and 2 ml each for the superficial peroneal nerve, saphenous nerve, and sural nerve.
  Other Names: Group 3
  Arms: 1% ropivacaine group

SUMMARY:
Peripheral nerve blocks are essential in ensuring effective regional anesthesia and postoperative analgesia in forefoot surgery for hallux valgus repair. Many factors influence the onset and duration of peripheral nerve blocks. In the advent of ultrasound-guided nerve blocks, the accuracy in administering LA has significantly improved, potentially reducing the required dosage, which is also associated with less risk for toxicity. However, the effect of the concentration of LA on the onset time and duration of ultrasound-guided ankle blocks for forefoot surgery has not yet been studied. This poses a clinically relevant dilemma regarding the necessity of administering lower or higher concentrations of ropivacaine to achieve a clinically relevant faster onset time and longer duration of an ankle block.

DETAILED DESCRIPTION:
This study aims to evaluate the differential effects of 0.25%, 0.5%, and 1% ropivacaine on the onset time and duration of ultrasound-guided ankle blocks in patients having forefoot surgery for anesthesia and postoperative analgesia. We hypothesize that the use of 1% ropivacaine for ultrasound guided ankle blocks will result in a significantly faster onset time and a longer sensory block duration, and thus analgesia, compared to the use of 0.25% and 0.5% ropivacaine in patients having forefoot surgery. The primary outcome is the difference in the duration of the sensory blocks. The secondary outcomes are the difference in onset time of the sensory block, motor function, the postoperative pain scores, opioid consumption, and proportion of failed blocks.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent
* Age 18 to 75 years, scheduled for elective forefoot surgery for hallux valgus repair under unilateral ankle block at ZOL Genk
* ASA physical I-II-III
* Able to ambulate (ability to walk independently, with or without assistive devices)
* Able to learn and perform study sensory and motor assessment by exhibiting sensitivity to pinprick, cold, and light touch (tested beforehand with pinprick/cold/ light touch sensation test) as the patient will have to perform these sensory and motor assessments by him/herself at home at postoperative day 0 to 2

Exclusion Criteria:

* Language barrier
* Preexisting lower extremity neuropathy
* Contraindications to ankle block (local infection, edema, burn, soft tissue trauma, or distorted anatomy with scarring in the area of block placement)
* Contraindications for use of NSAIDs
* Allergy to local anesthetics
* Uncontrolled anxiety, psychiatric or neurological disorder that might interfere with study assessment
* Weight below 50 kg based on a maximum dose of 3 mg/kg ropivacaine and a maximum dose of 150 mg ropivacaine.
* Preoperative use of opioids or gabapentin less than 3 days before surgery
* Contraindications for use of paracetamol
* Contraindications for use of tramadol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Duration | 48 hours
  The difference in sensory block duration across the different groups.

SECONDARY OUTCOMES:
Onset | 30 minutes
  The difference in sensory block onset across the different groups.
Motor function | 48 hours
  The difference in motor function across the different groups. The motor function will be evaluated with NRS during movement and at rest. The following scale will be used: 0 full strength, 1 ability to move but weakness experienced, 2 unable to move and no strength.
Pain scores | 48 hours
  The difference in postoperative pain scores across the different groups using a numeric rating scale from 0 being 'no pain' to 10 being 'worst pain imaginable'. The highest score (10) correlates with severe pain and thus worse outcome.
Opioid consumption | 48 hours
  The difference in opioid consumption across the different groups.
Proportion failed blocks | 48 hours
  The difference in the proportion of failed blocks across the different groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium